CLINICAL TRIAL: NCT06646731
Title: Ultrasound-guided Percutaneous Cryoneurolysis for Management of Chronic Painful Diabetic Neuropathy: A Randomized Sham-controlled Pilot Study
Brief Title: Cryoneurolysis for Painful Diabetic Neuropathy of the Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rodney Gabriel, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 811212
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Painful Diabetic Peripheral Neuropathy (PDPN)
Keywords: Cryoneurolysis; Diabetic Peripheral Neuropathy of the Foot; Chronic Pain; Ultrasound-Guided Percutaneous Cryoneurolysis
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study is a single-center, randomized, participant- and observer-masked, human-subjects, post-market clinical pilot study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (Active Comparator): For participants randomized to active treatment, the probe placed in the research participant will be triggered and the nitrous oxide passed through the probe and then back into the machine, and finally vented out from the console. This will result in a freeze-thaw cycle. This may be repeated, as necessary, to ensure the entire cross-section of each nerve is fully treated.
  Interventions: Device: cryoneurolysis
- Sham (Sham Comparator): Patients in this arm will also receive a diagnostic block with local anesthetic. If pain relief is satisfactory, the patients in this arm will undergo the procedure but the cryo probe will simply not be activated.
  Interventions: Device: sham cryoneurolysis

INTERVENTIONS:
Device: cryoneurolysis — Peripheral nerve cryoneurolysis of the foot
  Arms: Cryoneurolysis
Device: sham cryoneurolysis — a sham probe will be placed percutaneously proximal to target nerves. No cryoneurolysis will be given.
  Arms: Sham

SUMMARY:
The study is a single-center, randomized, participant- and observer-masked, human-subjects, post-market clinical pilot study to investigate the use of ultrasound-guided percutaneous cryoneurolysis to treat diabetic neuropathy of the foot. A prolonged nerve block may be provided by freezing the nerve using a technique called "cryoneurolysis". With cryoneurolysis and ultrasound machines, a small needle-like "probe" may be placed through anesthetized skin and guided to the target nerve to allow freezing. The procedure takes about 6 minutes for each nerve, involves little discomfort, has no systemic side effects, and cannot be misused or become addictive. Participants will be randomly allocated to one of two possible treatments groups: cryoneurolysis (experimental) or sham (control). The primary outcome measure is the change in pain on the neuropathic pain scale from baseline 1 month following the procedure.

DETAILED DESCRIPTION:
The study is a single-center, randomized, participant- and observer-masked, human-subjects, post-market clinical pilot study to investigate the use of ultrasound-guided percutaneous cryoneurolysis to treat diabetic neuropathy of the foot. A prolonged nerve block may be provided by freezing the nerve using a technique called "cryoneurolysis". With cryoneurolysis and ultrasound machines, a small needle-like "probe" may be placed through anesthetized skin and guided to the target nerve to allow freezing. The procedure takes about 6 minutes for each nerve, involves little discomfort, has no systemic side effects, and cannot be misused or become addictive. After 2-3 months, the nerve returns to normal functioning. Participants will be randomly allocated to one of two possible treatments groups: cryoneurolysis (experimental) or sham (control). The primary outcome measure is the change in pain on the neuropathic pain scale from baseline 1 month following the procedure.

Our objective is to investigate the therapeutic benefits of cryoneurolysis for research participants with painful diabetic neuropathy of the feet via a pilot study of 30 research participants. We hypothesize that ultrasound-guided cryoneurolysis of the superficial peroneal nerve will improve pain outcomes in research participants with painful diabetic neuropathy of the foot. The aims of this study will be to:

Primary Specific Aim. Demonstrate the potential efficacy of ultrasound-guided percutaneous cryoneurolysis of the superficial peroneal nerve, sural, distal saphenous, and/or deep peroneal nerve to treat painful diabetic neuropathy of the foot in reducing neuropathic pain 1 month after the procedure compared to baseline. This will be performed as a pilot study and executed as a randomized sham-controlled clinical trial of 30 subjects.

Hypothesis 1: Diabetic neuropathic pain intensity will be decreased relative to baseline 1 month following a cryoneurolysis procedure (as measured by the Neuropathic Pain Scale).

Secondary Specific Aim: To test the influence of a cryoanalgesia treatment as compared to sham/placebo on the long term measurements related to pain, quality of life, and analgesic usage.

Hypothesis 2a: Perception of well-being will be improved 1 month following one cryoneurolysis procedure (as measured with the Patient Global Impression of Change Scale).

Hypothesis 2b: Physical and emotional functioning will be improved relative to baseline 1 month following one cryoneurolysis procedure (as measured with the Interference Subscale of the Brief Pain Inventory).

Hypothesis 2c: Pain and opioid consumption will be reduced in the cryoneurolysis group compare to sham at multiple post-procedure time points, including 1 week, 1 month, 3 months, and 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* Research participants with diabetes mellitus and painful diabetic neuropathy of the foot (unilateral or bilateral)
* HgbA1c <10 (to avoid any increased risk of site infection)
* Adult patients of at least 18 years of age
* Experiencing at least moderate diabetic neuropathic pain in the foot - defined as 3 or higher on the numeric rating scale (NRS; 0-10, 0=no pain; 10=worse imaginable pain) - at least daily for the previous 2 months.

Exclusion Criteria:

* Diabetic neuropathy not in the distribution of the superficial peroneal nerve, sural nerve, deep peroneal, and/or distal saphenous nerve.
* Comorbidities that are contraindication to cryoneurolysis (e.g., Reynaud syndrome, cryoglobulinemia, cold urticaria)
* Allergy to local anesthetic
* Pregnancy
* Incarceration
* Inability to communicate to investigators due to lack of capacity
* Local infection in the foot/ankle where cryoneurolysis will be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 1 month
  Change in pain intensity compared to baseline due to diabetic neuropathy of the foot as measured by the score of the Neuropathic Pain Scale. The primary outcome will be at 1 month following the study procedure. The primary statistic will be comparing the median change in the neuropathic pain scale score between both cohorts.

SECONDARY OUTCOMES:
Perception of Well-Being | 1 month
  Perception of well-being will be improved 1 month following one cryoneurolysis procedure (as measured with the Patient Global Impression of Change Scale).
Physical and Emotional Functioning | 1 month
  Physical and emotional functioning will be improved relative to baseline 1 month following one cryoneurolysis procedure (as measured with the Interference Subscale of the Brief Pain Inventory).
Pain intensity - 1 month | 1 month
  Pain intensity as measured by Brief Pain Inventory
Pain Intensity - 1 week | 1 week
  Pain intensity as measured by Neuropathic Pain Scale and Brief Pain Inventory)
Pain Intensity - 3 months | 3 months
  Pain intensity as measured by the Brief Pain Inventory and Neuropathic Pain Scale
Pain Intensity - 6 months | 6 months
  Pain intensity as measured by the Brief Pain Inventory and Neuropathic Pain Scale
Opioid consumption - 1 week | 1 week
  opioid consumption as measured by the Quantitative Analgesic Questionnaire
Opioid consumption - 1 month | 1 month
  opioid consumption as measured by the Quantitative Analgesic Questionnaire
Opioid consumption - 3 months | 3 months
  opioid consumption as measured by the Quantitative Analgesic Questionnaire
Opioid consumption - 6 months | 6 months
  opioid consumption as measured by the Quantitative Analgesic Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided if we will share patient data with other researchers. Reasons for not sharing data would be related to patient confidentiality. Reasons to share data would be related to additional research analyses.

REFERENCES:
- [Background] Yoon JH, Grechushkin V, Chaudhry A, Bhattacharji P, Durkin B, Moore W. Cryoneurolysis in Patients with Refractory Chronic Peripheral Neuropathic Pain. J Vasc Interv Radiol. 2016 Feb;27(2):239-43. doi: 10.1016/j.jvir.2015.11.027. Epub 2015 Dec 17. PMID 26710969
- [Background] Jay GW, Barkin RL. Neuropathic pain: etiology, pathophysiology, mechanisms, and evaluations. Dis Mon. 2014 Jan;60(1):6-47. doi: 10.1016/j.disamonth.2013.12.001. No abstract available. PMID 24507705
- [Background] Gabriel RA, Seng EC, Curran BP, Winston P, Trescot AM, Filipovski I. A Narrative Review of Ultrasound-Guided and Landmark-based Percutaneous Cryoneurolysis for the Management of Acute and Chronic Pain. Curr Pain Headache Rep. 2024 Nov;28(11):1097-1104. doi: 10.1007/s11916-024-01281-z. Epub 2024 Jul 4. PMID 38963513
- [Background] Filipovski I, Gabriel RA, Kestenholz R. Ultrasound-Guided Cryoneurolysis for the Treatment of Painful Diabetic Neuropathy of the Foot: A Case Series. Cureus. 2024 Mar 16;16(3):e56267. doi: 10.7759/cureus.56267. eCollection 2024 Mar. PMID 38495961